CLINICAL TRIAL: NCT00533494
Title: The Effect of Patients' Participation in Improving Diabetes Care
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Soroka University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: sor166899ctil
Record Dates: First submitted 2007-09-20; First posted 2007-09-21 (Estimated); Last update posted 2007-11-14 (Estimated); Status verified 2003-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- B (Active Comparator): Feedback to physicians + reminder letters to patients
  Interventions: Behavioral: physician feedback (A)
- A (Active Comparator): Feedback information to physicians
  Interventions: Behavioral: physician feedback (A)

INTERVENTIONS:
Behavioral: physician feedback (A) — Feedback information to physicians

SUMMARY:
Despite the advent of efficacious medicines, there is a gap between ideal and actual care in the achievement of recommended outcomes among diabetic patients. The study enrolled 429 diabetic patients attending four HMO clinics in Israel, two in the northern region and two in the southern region. All clinics were randomly selected from all clinics affiliated with the Faculty of Health Sciences of the Ben Gurion University. The objective of the study was to compare the effects of a multi-component physician-patient intervention to physician feedback alone on a combined outcome of diabetes, blood pressure and serum lipids control. We hypothesized that in medical practices where physicians have received feedback on quality of care indicators, patients who received a letter encouraging them to discuss a list of important diabetes-related issues with their doctors, would experience better outcomes compared to patients who did no received such a letter.

ELIGIBILITY:
Inclusion Criteria:

* Known diabetic patients enrolled in the four primary care clinics
* Age 30 years and older.

Exclusion Criteria:

* Below age 30 years
* Type 1 diabetes
* Spoke neither Hebrew nor Russian
* Bedridden or confined to home.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-01; Study Completion 2003-09 (Actual)

PRIMARY OUTCOMES:
HbA1c, LDL, systolic blood pressure | Baseline and 1 year after 1-year intervention

CONTACTS AND LOCATIONS:
Overall Officials: Shimon Weitzman, MD, MPH, Study Chair — Department of Epidemiology- Faculty of Health Sciences-Ben Gurion University; Hava Tabenkin, MD, LLB, Principal Investigator — Department of Family Medicine, Afula - Clalit Health Services; Sheldon Greenfield, MD, Principal Investigator — Department of Medicine, School of Medicine,UCI; Sherrie H Kaplan, PhD, Principal Investigator — Department of Medicine, School of Medicine,ICI
Locations (1):
- Clalit Health Services, Beersheva, Afula, Migdal Haemek, Israel